CLINICAL TRIAL: NCT02339818
Title: Evaluation of the Effectiveness of Eliquis ® (Apixaban) Risk Minimization Tools in European Economic Area (EEA) Countries
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-365
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Stroke, Systemic Embolism, VTEt and VTEp
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HCPs: HCPs involved in using Eliquis (apixaban)
- Patients: Patients taking Eliquis for any of the three currently approved indications

SUMMARY:
The main purpose is to evaluate the effectiveness of the Eliquis® (apixaban) Prescriber Guide and Patient Alert Card in terms knowledge of the important identified risk of bleeding associated with Eliquis treatment communicated by the RM tools.

DETAILED DESCRIPTION:
Observational Model, Other- This is a non-interventional, cross-sectional study in the EEA involving representative samples of HCPs who treat patients with Eliquis, as well as patients treated with Eliquis. This study will be facilitated via web-based surveys used to evaluate the effectiveness of the Eliquis Prescribe Guide and Patient Alert Card as risk management tools.

Enrollment: 384 Health Care Professions (HCPs) and 192 Patients

Treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) and prevention of recurrent DVT and PE in adults (VTEt)

Prevention of VTE in adult patients knee replacement surgery (VTEp)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* HCP must have been involved in the treatment of at least one patient with Eliquis for any approved indication
* Patients must have taken Eliquis for any approved indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCPs will be considered for participation in the study if they prescribe/use Eliquis for any approved indications, including the following subgroups as appropriate for each country:
  * Cardiologists (including allied specialties, e.g. angiologists, electrophysiologists)
  * Non-cardiology specialists (e.g. internal medicine/hospital general medicine physicians, geriatricians/care of the elderly physicians, neurologists, hematologists, orthopedic surgeons)
  * General practitioners/internal medicine
  * Other HCPs (e.g. nurses, pharmacists)
  * Patients taking Eliquis for all three currently approved indications
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2015-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The proportions of HCPs using Eliquis and patients treated with Eliquis with knowledge of the important identified risk of bleeding associated with Eliquis treatment measured through web-based survey results | At the time of completion of a survey (approximately 6 to 12 months)

SECONDARY OUTCOMES:
The proportions of HCPs using Eliquis and patients treated with Eliquis who have received the Risk minimization (RM) tools measured through web-based survey results | At the time of completion of a survey (approximately 6 to 12 months)
The proportions of HCPs using Eliquis and patients treated with Eliquis who have utilized the RM tools, and the extent of tool usage measured through web-based survey results | At the time of completion of a survey (approximately 6 to 12 months)
The levels and distributions of behavior questionnaire results for HCPs and patients measured through web-based survey results | At the time of completion of a survey (approximately 6 to 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- [Derived] Mayall S, Kahlon R, Al-Dakkak I, Shen SW. Evaluating the Effectiveness of Apixaban Additional Risk Minimisation Measures Using Surveys in Europe. Pharmaceut Med. 2021 Mar;35(2):123-135. doi: 10.1007/s40290-021-00380-1. Epub 2021 Mar 4. PMID 33660230
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx